CLINICAL TRIAL: NCT01504451
Title: Left Atrial Ablation of Paroxysmal Atrial Fibrillation With Implantable Loop Recorder Follow Up Study 2
Brief Title: Left Atrial Ablation of Paroxysmal Atrial Fibrillation With Implantable Loop Recorder Follow Up Study: The LAAPITUP 2 Study
Acronym: LAAPITUP 2
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Neil Sulke (Other)
Responsible Party: Sponsor-Investigator, Neil Sulke, Consultant Cardiologist, Eastbourne General Hospital
Organization: Eastbourne General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LAAPITUP 2
Record Dates: First submitted 2011-12-30; First posted 2012-01-05 (Estimated); Last update posted 2014-06-26 (Estimated); Status verified 2014-06

CONDITIONS: Paroxysmal Atrial Fibrillation
Keywords: Atrial fibrillation; Ablation; Implantable loop recorder
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Biosense Webster ablation (Active Comparator): Biosense Webster irrigated multi-electrode phased radiofrequency AF ablation
  Interventions: Device: ILR insertion; Procedure: AF ablation
- Surgical ablation (Active Comparator): Minimally invasive thoracoscopic surgical AF ablation
  Interventions: Device: ILR insertion; Procedure: AF ablation
- Medtronic ablation (Active Comparator): Medtronic multi-electrode phased radiofrequency AF ablation
  Interventions: Device: ILR insertion; Procedure: AF ablation

INTERVENTIONS:
Device: ILR insertion — Insertion of implantable loop recorder
Procedure: AF ablation — AF ablation

SUMMARY:
This study is designed to compare three different techniques in ablation of paroxysmal atrial fibrillation. Namely, the Medtronic multi-electrode phased radiofrequency ablation system, the Biosense Webster irrigated multi-electrode phased radiofrequency ablation system, and minimally invasive thoracoscopic surgical ablation. The study hypothesis is that surgical and Biosense Webster ablation are non-inferior to Medtronic ablation.

DETAILED DESCRIPTION:
A target of 75 participants will be randomised 1:1:1 to one of the three treatment arms. Each participant will have an implantable loop recorder (ILR) prior to ablation in order to assess AF burden. After ablation, each participant will be followed up for a year. The ILR will be used to assess reduction in AF burden.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic paroxysmal AF suitable for AF ablation
* Age > 18 years old
* Informed consent to participate in this study.

Exclusion Criteria:

* Pre-existing ILRs or permanent pacemakers that do not allow for continuous monitoring for AF occurrence, or are not MRI-safe.
* Unable to undergo general anaesthesia for AF ablation.
* Previous cardiac surgery, such as coronary artery bypass grafting or valvular surgery.
* Scheduled for elective cardiac surgery, such as coronary artery bypass grafting or valvular surgery.
* Previous thoracic surgery.
* Participation in a conflicting study.
* Potential participants who are mentally incapacitated and cannot consent or comply with follow-up
* Pregnancy
* Other cardiac rhythm disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2012-04; Primary Completion 2015-04 (Estimated); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
AF burden | 12 months after ablation
  Total proportion of time spent in AF as assessed by ILR

SECONDARY OUTCOMES:
Time to AF recurrence | Up to one year
  Time to recurrence of any AF after ablation
Time to first symptomatic AF recurrence | Up to one year
  Time to first symptomatic AF recurrence as assessed by ILR.
Change in QoL measures | 12 months after ablation
  Change in Quality of Life measures assessed by questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Neil Sulke, MD, Principal Investigator — Eastbourne General Hospital; Stephen S Furniss, MD, Principal Investigator — Eastbourne General Hospital
Locations (2):
- United Kingdom (2):
  - Eastbourne General Hospital, Eastbourne, E Sussex
  - Royal Sussex County Hospital, Brighton, Sussex

REFERENCES:
- [Derived] Sugihara C, Furniss S, Hyde J, Lewis M, Sulke N. Results of the first investigator-initiated randomized clinical trial of nMARQTM, PVACTM, and thoracoscopic ablation for paroxysmal atrial fibrillation. Europace. 2018 Nov 1;20(FI_3):f384-f391. doi: 10.1093/europace/eux267. PMID 29092038